CLINICAL TRIAL: NCT06707805
Title: Effects of Lumber Sustained Natural Apophyseal Glides on Lower Cross Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: REC/MS-PT/01879 Amreen Shabbir
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Lower Cross Syndrome
Keywords: pain; lumber SNGS
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lumber SNAGS (Experimental): A sustained natural apophyseal glide (SNAG) is a mobilization technique commonly used in the treatment of painful movement restrictions of the spine.Studing the effect of Lumber SNAGs in lower cross syndrome hold significance due to its potential to correct pain, hypomobility and biomechanical changes i.e hyperlordotic curve and anterior pelvic tilting caused by lower cross syndrome
  Interventions: Other: lumber SNAGS
- Conventional group (Other): Exercises ,Tens and hotpack
  Interventions: Other: Traditional Physical therapy

INTERVENTIONS:
Other: Traditional Physical therapy — Conventional treatment protocol including moist Heating pad for low back pain for 15 minutes. TENS for pain for 10 minutes. Stretchings of tight muscles would be 1 set of 5-7 reps with 5 sec. hold 3 times a week. Strengthing of weak muscles would be 2-3 times a weak with 10-15 reps.Stretching protocol will be followed for Iliopsoas and erector spinae muscles. Strengthening protocol will be followed for weak abdominals and Gluteus maximus muscles
  Arms: Conventional group
Other: lumber SNAGS — : Lumber mobilizations with conventional treatment protocol.
  * Lumber Mulligan(SNAGs) technique
  * Technique applied at L4-L5, L5-S1 level.
  * Techniques applied for flexion ,extension, side bending and rotation 6 to 8 cycles per session
  Arms: lumber SNAGS

SUMMARY:
A sustained natural apophyseal glide (SNAG) is a mobilization technique commonly used in the treatment of painful movement restrictions of the spine.Studing the effect of Lumber SNAGs in lower cross syndrome hold significance due to its potential to correct pain, hypomobility and biomechanical changes i.e hyperlordotic curve and anterior pelvic tilting caused by lower cross syndrome. The specific muscle imbalance seen in PCS gives rise to specific joint dysfunction, particularly in the L4-L5 and L5-S1 segment of the vertebral column. Over time, this causes stress at the L5-S1 segment of the vertebral column leading to pain and irritation in the lower back Lumber SNAGs encourage improvement of these repositioning error, posture, alleviate discomfort and enhance overall functioning. This research aims to offer patients a noninvasive and personalized approach to managing LCS, ultimately contributing to their overall well-being and movement quality

DETAILED DESCRIPTION:
A sustained natural apophyseal glide (SNAG) is a mobilization technique commonly used in the treatment of painful movement restrictions of the spine.Studing the effect of Lumber SNAGs in lower cross syndrome hold significance due to its potential to correct pain, hypomobility and biomechanical changes i.e hyperlordotic curve and anterior pelvic tilting caused by lower cross syndrome. The specific muscle imbalance seen in PCS gives rise to specific joint dysfunction, particularly in the L4-L5 and L5-S1 segment of the vertebral column. Over time, this causes stress at the L5-S1 segment of the vertebral column leading to pain and irritation in the lower back Lumber SNAGs encourage improvement of these repositioning error, posture, eleviate discomfort and enhance overall functioning. This research aims to offer patients a noninvasive and personalized approach to managing LCS, ultimately contributing to their overall well-being and movement quality The significance of this study lies in it's potential to improve the health and wellbeing of adults have pain and hypomobility due to lower cross syndrome.By identifying an effective physical therapy intervention for correcting pain and hypomobility , this study provide valueable insight for clinicians in develping effective treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 50 years.
* Both genders
* Patient came with the complain of low back pain.
* Participants had to present with pain and hypomobility due to lower cross syndrome
* Participants had to meet the criteria for lower cross syndrome indicating tight hip flexors and erector spinae along with weak abdominals and glutei muscles
* Participants with hyperlordotic curve due to lower cross syndrome
* Participants presenting with anterior pelvic tilting greater than angle >7-10 degrees
* Willing to provide informed consent to participate in study

Exclusion Criteria:Participants contraindicated to spinal manipulation

* Musculoskeletal pathologies affecting the lower back, pelvis, hips, or lower extremities (e.g., herniated disc, lumbar radiculopathy, lumbar stenosis, hip labral tear).
* Participants who had undergone any lumber or pelvic surgery, as it will affect sacroiliac joint mechanics.
* Generalized inflammatory or infective connective tissue disorder
* Pregnancy

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Oswestry disability index | from baseline to 4th week
  The Oswestry Low Back Pain Disability Questionnaire is an adequate apparatus used to measure disability caused by low back pain in the general population. The questionnaire examines the level of disability in 10 everyday activities of daily living. Each item consist of 6 statements which are scored from 0 to 5. With 0 indicating the least disability and 5 the greatest then the total score is calculated as a percentage, with 0% indicating no disability and 100% indicating the highest level of disability.

SECONDARY OUTCOMES:
Numeric pain rating sacle | from baseline to 4th week
  The Numerical Rating Scale (Appendix G) is one of the most commonly used tools to measure pain intensity in both clinical and research settings. The Numerical Rating Scale is an 11-point scale that consists of numbers from 0 to 10, 0 signifies "no pain" and 10 signifies "worst imaginable pain"
Lumber Range of motion | AT baseline and 3rd week
  to test hypomobility in Lumber Spine with the help of Inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Asmar Fatima, MS OMPT, Principal Investigator — Riphah International University
Locations (1):
- Orthopaedic hospital, Kotli, Azad Kashmir, Pakistan

IPD SHARING:
Plan to Share IPD: No